CLINICAL TRIAL: NCT04031404
Title: Modulation of Motor Cortex Excitability by Glucose Administration
Brief Title: Glucose and Non-Invasive Brain Stimulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 19-1451
Record Dates: First submitted 2019-07-18; First posted 2019-07-24 (Actual); Results first posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-08

CONDITIONS: Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The researcher that interacts with the subject will not know whether the subject consumed the glucose drink or the placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Glucose drink followed by placebo (Experimental): Participants will consume the glucose drink at session 1, then they will consume the placebo (water) at session 2.
  Interventions: Device: Single-pulse TMS
- Placebo followed by glucose drink (Experimental): Participants will consume the placebo (water) at session 1, then they will consume the glucose drink at session 2.
  Interventions: Device: Single-pulse TMS

INTERVENTIONS:
Device: Single-pulse TMS — Single-pulse transcranial magnetic stimulation (TMS) on the motor cortex will lead to a twitch in the target muscle and evoke a motor-evoked potential (MEP) measured by electromyography (EMG).
  Other Names: MagPro X100

SUMMARY:
Purpose: In this study, the investigators will delineate how brain network dynamics are modulated by experimentally induced elevated blood glucose levels and examine how glucose levels gate neuronal excitability measured by the response to TMS.

Participants: Participants must be between the ages of 18 and 65 with no known diabetes, no known adverse reaction to finger prick blood draw, and no known neurological or psychiatric illness. Participants must have a body-mass index less than 30.

Procedures: Participants will consume either a drink that contains 75 g of glucose or a placebo, and their response to TMS will be measured to examine the effect of glucose on motor cortex excitability.

DETAILED DESCRIPTION:
This study will be a placebo-controlled study that investigates brain function with both electroencephalography (EEG) and TMS. On each study visit, a drink (either glucose drink or water) is administered after baseline assessment of fasting glucose. Changes in brain activity and excitability will be measured with resting-state EEG. Periodic high-density EEG of resting-state brain activity and activity during a working memory task will be performed before the administration of the drink, immediately after the administration of the drink, as well as 30 minutes, 60 minutes, 120 minutes, 150 minutes, and 180 minutes after the administration of the drink. The spectral content of the EEG signal will be investigated to identify the relative presence of cortical oscillations. Primarily, there will be a focus on theta (4-8 Hz) and alpha (8-12 Hz) oscillations.

Previous literature indicates that theta and alpha oscillations represent an engaged and disengaged cortical state, respectively [1]. Alpha and theta oscillations are implicated in cognitive function and are altered in depression. Therefore, this study aims to identify a decrease in frontal theta oscillations and an increase in left frontal alpha oscillations, two defining features of impaired top-down control and mood regulation, in response to the glucose drink contrasted with the response to the placebo.

The study will also examine how glucose levels gate neuronal excitability measured by the response to TMS. Cortical excitability will be measured by applying TMS pulses to the motor cortex and measuring the response in the form of a motor evoked potential by electromyography (EMG). TMS will be applied before the administration of the drink, immediately after the administration of the drink, as well as 30 minutes, 60 minutes, 120 minutes, 150 minutes, and 180 minutes after the administration of the drink. Changes in blood glucose will be monitored over this time interval as well.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* BMI <30
* Free of major neurological conditions and diabetes

Exclusion Criteria:

* Diabetes
* Adverse reaction to finger prick blood draw
* Known neurological or psychiatric illness
* Prior brain surgery
* Any brain devices/implants, including cochlear implants and aneurysm clips
* Cardiac pacemaker
* Any other implanted electronic device
* History of current traumatic brain injury
* Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, Principal Investigator — Carolina Center for Neurostimulation
Locations (1):
- UNC Medical School Wing C, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication.
Access Criteria: IRB, IEC, or REB approval, as applicable, and execution of a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Stitt I, Zhou ZC, Radtke-Schuller S, Frohlich F. Arousal dependent modulation of thalamo-cortical functional interaction. Nat Commun. 2018 Jun 25;9(1):2455. doi: 10.1038/s41467-018-04785-6. PMID 29941957

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Glucose Drink Followed by Placebo | Placebo Followed by Glucose Drink
Started (Randomized) | 10 | 13
Completed | 8 | 8
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Did not meet full inclusion/exclusion. | 2 | 4
Period: Pre-randomization
Arm/Group | Glucose Drink Followed by Placebo | Placebo Followed by Glucose Drink
Started | 8 | 8
Completed | 6 | 5
Not Completed | 2 | 3
Not completed — Withdrawn for COVID19 precautions | 1 | 3
Not completed — Disqualified by TMS safety screening | 1 | 0
Period: First Drink Visit
Arm/Group | Glucose Drink Followed by Placebo | Placebo Followed by Glucose Drink
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout (5 Day Min)
Arm/Group | Glucose Drink Followed by Placebo | Placebo Followed by Glucose Drink
Started | 6 | 5
Completed | 5 | 5
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Second Drink Visit
Arm/Group | Glucose Drink Followed by Placebo | Placebo Followed by Glucose Drink
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants will consume the glucose drink at session 1, then they will consume the placebo (water) at session 2, or vice versa.
  Single-pulse TMS: Single-pulse transcranial magnetic stimulation (TMS) on the motor cortex will lead to a twitch in the target muscle and evoke a motor-evoked potential (MEP) measured by electromyography (EMG).
Arm/Group | All Participants
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.64 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 13
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Motor Evoked Potential (MEP)
Description: Change in MEP over time to indicate changes in motor cortex excitability
Time Frame: Measurements will be taken before the administration of the drink, as well as 0, 30, 60, 120, and 180 minutes after the administration of the drink.
Population: From the 10 participants who completed, 3 were excluded from the analysis due to technical reasons. Two participants had to end their glucose visits early due to scheduling conflicts. The reported N below is adjusted where appropriate.
Measure: Mean (Standard Error); unit: log10(Post uV/Baseline uV)
Groups:
- MEP After Glucose Drink: Participants receive TMS to motor cortex following consumption of a 75 g glucose drink (~300 mL).
- MEP After Placebo Drink: Participants receive TMS to motor cortex following consumption of a water control (~300 mL).
Arm/Group | MEP After Glucose Drink | MEP After Placebo Drink
Number analyzed (Participants) | 7 | 7
log10(Post uV/Baseline uV)
  MEP change (0 min vs pre-drink) | 0.14 (0.15) | -0.25 (0.07)
  MEP change (30 min vs pre-drink) | -0.02 (0.19) | -0.12 (0.11)
  MEP change (60 min vs pre-drink) | -0.08 (0.14) | -0.33 (0.10)
  MEP change (120 min vs pre-drink) | -0.05 (0.16) | -0.25 (0.09)
  MEP change (180 min vs pre-drink): number analyzed (Participants) | 5 | 7
  MEP change (180 min vs pre-drink) | -0.21 (0.18) | -0.18 (0.10)

2. Primary Outcome: TMS Evoked Potential (TEP)
Description: The TMS Evoked Potential (TEP) is the difference in microvolts from 25 milliseconds after a TMS pulse versus pre-TMS such that greater values indicate greater motor cortex excitability. The measure of the change in TEP over time since either glucose or water was consumed approximates a z-distribution with a range of -20 to 20 with central distribution measures of zero. TEPs were source localized and reported using a pseudo-neural activity index (PNAI) expressing source activation in relation to pre-TMS pulse trial baseline. The difference in the source peaks corresponding to the early P25 component have been reported as differences from baseline. Higher values indicate greater cortical excitation, consistent with the study hypothesis.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: z-score
Groups:
- Source-localized TEP After Glucose Drink: Participants receive TMS to motor cortex following consumption of a 75 g glucose drink (~300 mL).
- Source-localized TEP After Placebo Drink: Participants receive TMS to motor cortex following consumption of a water control (~300 mL).
Arm/Group | Source-localized TEP After Glucose Drink | Source-localized TEP After Placebo Drink
Number analyzed (Participants) | 7 | 7
z-score
  TEP change (P25: 0 min vs pre-drink) | -0.04 (0.08) | 0.28 (0.16)
  TEP change (P25: 30 min vs pre-drink) | -0.11 (0.11) | 0.024 (0.05)
  TEP change (P25: 60 min vs pre-drink) | -0.16 (0.11) | 0.30 (0.06)
  TEP change (P25: 120 min vs pre-drink) | -0.16 (0.12) | 0.24 (0.07)
  TEP change (P25: 180 min vs pre-drink): number analyzed (Participants) | 5 | 7
  TEP change (P25: 180 min vs pre-drink) | 0.08 (0.08) | 0.02 (0.15)

3. Secondary Outcome: EEG Measure of Alpha Asymmetry Oscillations
Description: Electroencephalography will be used to measure the change in lateralized alpha asymmetry (10-12 Hz electrical activity) over time
Time Frame: as for outcome 1
Population: From the 10 participants who completed, one was excluded from the analysis due to technical reasons. Two participants had to end their glucose visits early due to scheduling conflicts. The reported N below is adjusted where appropriate.
Measure: Mean (Standard Error); unit: 10*log10(Right Alpha/Left Alpha) (uV)
Groups:
- Alpha Asymmetry After Glucose Drink; Alpha Asymmetry After Placebo Drink: Participants complete a resting state EEG recording following consumption of a 75 g glucose drink (~300 mL).
Arm/Group | Alpha Asymmetry After Glucose Drink | Alpha Asymmetry After Placebo Drink
Number analyzed (Participants) | 9 | 9
10*log10(Right Alpha/Left Alpha) (uV)
  Alpha Asymm. Change (0 min vs Baseline) | 0.15 (0.15) | 0.59 (0.45)
  Alpha Asymm. Change (30 min vs Baseline) | -0.01 (0.20) | 0.42 (0.42)
  Alpha Asymm. Change (60 min vs Baseline) | 0.14 (0.22) | 0.19 (0.25)
  Alpha Asymm. Change (120 min vs Baseline) | 0.18 (0.22) | 0.33 (0.22)
  Alpha Asymm. Change (180 min vs Baseline): number analyzed (Participants) | 7 | 9
  Alpha Asymm. Change (180 min vs Baseline) | 0.18 (0.33) | 0.28 (0.33)

4. Secondary Outcome: EEG Measure of Frontal Midline Theta Oscillations
Description: Electroencephalography will be used to measure the change in frontal midline theta power (5-8 Hz electrical activity) over time
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Error); unit: 10*log10(Post uV/Baseline uV)
Groups:
- Midline Frontal Theta Oscillations After Glucose Drink; Midline Frontal Theta Oscillations After Placebo Drink: Participants complete a resting state EEG recording following consumption of a 75 g glucose drink (~300 mL).
Arm/Group | Midline Frontal Theta Oscillations After Glucose Drink | Midline Frontal Theta Oscillations After Placebo Drink
Number analyzed (Participants) | 9 | 9
10*log10(Post uV/Baseline uV)
  Theta Power Change (0 min vs Baseline) | 0.12 (0.34) | 0.33 (0.28)
  Theta Power Change (30 min vs Baseline) | 0.56 (0.25) | 0.57 (0.27)
  Theta Power Change (60 min vs Baseline) | 0.94 (0.29) | 1.15 (0.32)
  Theta Power Change (120 min vs Baseline) | 0.36 (0.26) | 1.21 (0.45)
  Theta Power Change (180 min vs Baseline): number analyzed (Participants) | 7 | 9
  Theta Power Change (180 min vs Baseline) | 1.48 (0.32) | 0.72 (0.34)

5. Secondary Outcome: Working Memory Task Accuracy
Description: This outcome will analyze the change in accuracy in a computerized working memory task over time. During the task, subjects will be presented with an array of colored squares. Then, they will need to hold this array in mind during a delay period. Finally, participants will be tested on their memory of the array by responding whether a presented color is the same or different as the corresponding square in the first array. Participants' accuracy will be expressed as the percentage of correct responses (from 0% correct responses to 100% correct responses). An accuracy rate of 50% indicates that the participant is performing at the same accuracy level as random chance.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Ratio of correct responses
Groups:
- Working Memory Accuracy After Glucose Drink: Participants complete a working memory task following consumption of a 75 g glucose drink (~300 mL).
- Midline Frontal Theta Oscillations After Placebo Drink: Participants complete a working memory task recording following consumption of a 75 g glucose drink (~300 mL).
Arm/Group | Working Memory Accuracy After Glucose Drink | Midline Frontal Theta Oscillations After Placebo Drink
Number analyzed (Participants) | 9 | 9
Ratio of correct responses
  WM Accuracy (0 min vs Baseline) | 1.02 (0.03) | 0.97 (0.03)
  WM Accuracy (30 min vs Baseline) | 1.02 (0.02) | 0.99 (0.03)
  WM Accuracy (60 min vs Baseline) | 1.06 (0.02) | 1.01 (0.03)
  WM Accuracy (120 min vs Baseline) | 1.05 (0.03) | 1.02 (0.03)
  WM Accuracy (180 min vs Baseline): number analyzed (Participants) | 7 | 9
  WM Accuracy (180 min vs Baseline) | 1.03 (0.03) | 1.03 (0.03)

ADVERSE EVENTS:
Time Frame: Up to 2 months per participant
Groups:
- TMS-EEG After Glucose Drink: Participants receive TMS to motor cortex following consumption of a 75 g glucose drink (~300 mL).
  During every session, participants receive single pulse TMS to the motor cortex, and complete EEG recordings and a working memory task at several time points.
- TMS-EEG After Placebo Drink: Participants receive TMS to motor cortex following consumption of a water control drink (~300 mL).
  During every session, participants receive single pulse TMS to the motor cortex, and complete EEG recordings and a working memory task at several time points.
Arm/Group | TMS-EEG After Glucose Drink | TMS-EEG After Placebo Drink
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 10/11 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS-EEG After Glucose Drink (N=11) | TMS-EEG After Placebo Drink (N=10)
Ringing or buzzing noise (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Dizziness (General disorders) | 3 (3) | 1 (1)
Sleepiness (General disorders) | 8 (8) | 5 (5)
Trouble concentrating (General disorders) | 4 (4) | 2 (2)
Headache (General disorders) | 5 (5) | 3 (3)
Itching (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Local redness (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Tingling (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Worsening mood (Psychiatric disorders) | 5 (5) | 2 (2)
Flickering lights (General disorders) | 0 (0) | 0 (0)
Burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Neck pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The end sample sizes are lower than intended as the trial was ended early due to COVID-19-related research drawdowns. Technical limitations in the Electroencephalogram (EEG) and Transcranial Magnetic Stimulation (TMS) data collection resulted in N=1 and N=3 dataset to be excluded from final analyses, respectively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT04031404/Prot_SAP_000.pdf